CLINICAL TRIAL: NCT06791876
Title: 'Nurture and Play' - a Randomized Controlled Pilot Study of a Perinatal Intervention to Strengthen Parenting Among Women with Psychosocial Vulnerabilities and Their Partners.
Brief Title: 'Nurture and Play' - a Pilot Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Clinical Research and Prevention (Network)
Collaborators: University of Copenhagen (Other); Slagelse Sygehus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-24058743
Record Dates: First submitted 2025-01-14; First posted 2025-01-24 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2024-11

CONDITIONS: Depression, Anxiety; Intervention; Randomized Controlled Study
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The parents who agree to participate in the study will be randomly assigned in a 1:1 ratio to either the intervention, Nurture and Play, or the control group, using random permuted block randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The intervention group - The Nurture and Play group program (Experimental): In addition to care-as-usual, the intervention group will be offered to participate in the NnP adapted to include partners. The intervention consists of 11 group sessions (4 prenatal and 11 postnatal sessions) and will be provided to parents in the intervention group from around pregnancy week 26 until the child is around seven months old. Each group will consist of four to five mothers/couples. The intervention will be delivered by midwives and health nurses who will receive training in conducting the program. The training for the professionals will be delivered by the Finish group which has developed the program and consists of four days of training - two days introductory and two days of training that will be given after some practice with the program.
  Interventions: Behavioral: Nurture and Play (NnP)
- The control group - Care as Usual (No Intervention): The control group are offered a basic package of antenatal care consisting of three consultations with their general practitioner, two ultrasound examinations, and four to seven consultations with midwives depending on parity. Postnatal examinations of the infant are performed regularly by the health nurse in the infant's home. During the child's first year, the health nurse examines the infant at least twice within the first three weeks after birth, at two months, at four months (for first-time mothers) and again at eight months. Extra counselling home visits to vulnerable families after the infant is born are provided by health nurses in all municipalities with the number and content depending on families' specific needs.

INTERVENTIONS:
Behavioral: Nurture and Play (NnP) — The NnP group Intervention is a group-based, manualized parenting intervention initiated during pregnancy and continued into the postnatal period until infant age seven months. The program is designed to enhance parenting abilities focusing on three domains: Emotional availability, parental reflective functioning, and the ability to regulate own emotions. During NnP, the parents are supported in enhancing their emotional availability through caring and playing activities.
  The intervention has been developed in Finland by Dr. Saara Salo and colleagues and tested in a randomized controlled trial among pregnant women with depression and it is now being implemented in Finland. The results from the study showed that mothers in the intervention group showed more emotional availability and higher levels of reflective functioning and experienced fewer depressive symptoms compared to mothers in the control group.
  Arms: The intervention group - The Nurture and Play group program

SUMMARY:
The aim of this randomised controlled pilot study is to evaluate the feasibility of the Nurture and Play (NnP) offered to a Danish population of psychosocial vulnerable pregnant women and their partners.

More specifically the objectives of the study are to:

* Test the feasibility of the NnP including both parents
* Evaluate the recruitment procedure, the adherence as well as the participant's and professional´s experience of the intervention
* Evaluate the collaboration between the hospitals and the municipalities.

The study consists of:

1. A randomized controlled pilot study (n=20 women/couples) carried out according to the Standard Protocol Items: Recommendations for Interventional Trials SPIRIT statement for clinical trials. The parents who agree to participate in the study will be randomly assigned in a 1:1 ratio to either the intervention or the control group. In addition to care-as-usual, the intervention group will be offered to participate in the NnP adapted to include partners. The intervention consists of 11 group sessions (4 perinatal and 7 postnatal sessions) and will be provided to the parents in the intervention group from around 26 weeks gestation until the baby is around seven months old. Each group session will be led by a midwife and a health nurse and will consist of four to five mothers/couples.
2. A qualitative descriptive interview study aiming to evaluate the participants' and professionals´ experience of the intervention.

Data will be collected through:

* Online Questionnaires.
* Interviews.
* Videotaped settings.

DETAILED DESCRIPTION:
Protocol

Title 'Nurture and Play' - a randomized controlled pilot study of a perinatal intervention to strengthen parenting among women with psychosocial vulnerabilities and their partners.

The aim of this randomised controlled pilot study is to evaluate the feasibility of the Nurture and Play (NnP) offered to a Danish population of psychosocial vulnerable pregnant women and their partners.

More specifically the objectives of the study are to:

* Test the feasibility of the NnP including both parents
* Evaluate the recruitment procedure, the adherence as well as the participant's and professional´s experience of the intervention
* Evaluate the collaboration between the hospitals and the municipalities.

The investigators hypothesize that the intervention can strengthen the quality of parent-infant interactions, enhance parental reflective functioning, and improve parental mental well-being. Further, the investigators expect that providing the intervention will strengthen the collaboration between hospitals and municipalities and build an early foundation for a fruitful and secure partnership between future parents and the health and social care system.

Conducting a pilot study provides the opportunity to test the trial in a smaller scale before initiating the full-scale and thereby strengthen the trial.

Background The foundation of children´s physical, mental, and cognitive development is established before birth and is affected by social and psychological risk factors connected to the parents. Meta-analyses have documented that the well-being of the mother during pregnancy both directly and indirectly affects the fetus and the child´s later development. As such, prenatal psychological stress and depression in pregnant women increase the risk of premature birth and low birth weight. Additionally, untreated stress and depression during pregnancy is indirectly related to later developmental problems in the child such as altered stress response, attention deficit hyperactive disorder, depression, and anxiety, e.g. by affecting the mother's parenting skills. Finally, studies have shown that maternal well-being during pregnancy affects the pregnant woman´s emotional involvement with her unborn infant - a prerequisite for later parenting skills. Around 10-15% have symptoms of depression during pregnancy, 15% of anxiety, and the prevalence of antenatal mental health problems is increasing.

A recent systematic review and meta-analysis found that perinatal interventions for women with antenatal depression can decrease the offspring's risk of psychopathology. Core components of effective perinatal interventions for infants of mothers psychosocial vulnerabilities are: Facilitation of positive mother-infant interactions, helping mothers to understand the infant´s perspective, and where applicable the use of video-feedback on parent-infant interactions. Existing perinatal care for pregnant women with psychosocial vulnerabilities in Denmark consists of an interdisciplinary and intersectoral collaboration between midwives, obstetricians, psychiatrists, primary sector health nurses, and general practitioners as well as social workers and family therapists. However, despite the international evidence regarding the effect of perinatal interventions to support parenting, such interventions are not part of the existing Danish perinatal program for women with psychosocial vulnerabilities. In line with this, qualitative interviews conducted by this research group with families with psychosocial vulnerabilities focusing on their need for care and support as a preparation for this project, highlighted the need for 1) more integration of the care provided by midwives and the municipalities, 2) more support for their mental well-being and 3) support to the partners.

The NnP group Intervention (in Danish: 'Omsorg og leg' - for dig og din baby) is a group-based, manualized parenting intervention initiated during pregnancy and continued into the postnatal period until infant age seven months. The program is designed to enhance parenting abilities focusing on three domains: Emotional availability, parental reflective functioning, and the ability to regulate own emotions. Emotional availability refers to the parent´s ability to read and respond appropriate to infant's emotional signals, similar to the attachment concept of parental sensitivity. During NnP, the parents are supported in enhancing their emotional availability through caring and playing activities. These include prenatal activities like singing and playing musical instruments for the future child and postnatal activities such as baby massage and interactive playing, like peekaboo. These activities are designed to enhance an emotional loving contact with the future child through physical contact and reciprocity and after birth shared attention with the child. In addition, each session also contains discussions about a particular theme chosen to activate parents´ reflective functioning, such as thoughts and feelings related to pregnancy and parenthood, memories of their childhood, expectations about their child, prior experiences with pregnancy and parenthood and hopes for own and their child future. Finally, each session contains a psycho-educative component focusing on strategies for regulating own emotions. The intervention has been developed in Finland by Dr. Saara Salo and colleagues and tested in a randomized controlled trial among pregnant women with depression and it is now being implemented in Finland. The results from the study showed that mothers in the intervention group showed more emotional availability and higher levels of reflective functioning and experienced fewer depressive symptoms compared to mothers in the control group. The Nurture and Play program have not been evaluated in a Danish context, which is relevant due to potential differences in the characteristics of the study population and the antenatal care program.

1. Heckman JJ. Skill formation and the economics of investing in disadvantaged children. Science. 2006;312(5782):1900-2.
2. Grote NK, Bridge JA, Gavin AR, Melville JL, Iyengar S, Katon WJ. A Meta-analysis of Depression During Pregnancy and the Risk of Preterm Birth, Low Birth Weight, and Intrauterine Growth Restriction. Archives of General Psychiatry. 2010;67(10):1012-24.
3. Grigoriadis S, VonderPorten EH, Mamisashvili L, Tomlinson G, Dennis C-L, Koren G, et al. The impact of maternal depression during pregnancy on perinatal outcomes: a systematic review and meta-analysis. The Journal of clinical psychiatry. 2013;74(4):0-.
4. Szegda K, Markenson G, Bertone-Johnson ER, Chasan-Taber L. Depression during pregnancy: a risk factor for adverse neonatal outcomes? A critical review of the literature. The Journal of Maternal-Fetal & Neonatal Medicine. 2014;27(9):960-7.
5. Graignic-Philippe R, Dayan J, Chokron S, Jacquet A, Tordjman S. Effects of prenatal stress on fetal and child development: a critical literature review. Neuroscience & biobehavioral reviews. 2014;43:137-62.
6. Waters CS, Hay DF, Simmonds JR, van Goozen SH. Antenatal depression and children's developmental outcomes: potential mechanisms and treatment options. European child & adolescent psychiatry. 2014;23(10):957-71.
7. Stein A, Pearson RM, Goodman SH, Rapa E, Rahman A, McCallum M, et al. Effects of perinatal mental disorders on the fetus and child. Lancet. 2014;384(9956):1800-19.
8. Pearson RM, Evans J, Kounali D, Lewis G, Heron J, Ramchandani PG, et al. Maternal depression during pregnancy and the postnatal period: risks and possible mechanisms for offspring depression at age 18 years. JAMA psychiatry. 2013;70(12):1312-9.
9. Foley S, Hughes C. Great expectations? Do mothers' and fathers' prenatal thoughts and feelings about the infant predict parent-infant interaction quality? A meta-analytic review. Developmental Review. 2018;48:40-54.
10. Antenatal and postnatal mental health: The NICE guideline on clinical management and service guidance. NICE guideline CG45. London: The Royal College of Psychiatrists; 2007.
11. Goodman SH, Cullum KA, Dimidjian S, River LM, Kim CY. Opening windows of opportunities: Evidence for interventions to prevent or treat depression in pregnant women being associated with changes in offspring's developmental trajectories of psychopathology risk. Development and Psychopathology. 2018;30(3):1179-96.
12. Newton K, Taylor Buck E, Weich S, Uttley L. A review and analysis of the components of potentially effective perinatal mental health interventions for infant development and mother-infant relationship outcomes. Development and Psychopathology. 2020:1-18.
13. Salo SJ, Lampi H. Nurture and Play Intervention for Groups. . 2019.
14. Biringen Z. Emotional availability: Conceptualization and research findings. American Journal of Orthopsychiatry. 2000;70(1):104-14.
15. Ainsworth MDS, Blehar MC, Waters E, Wall S. Patterns of Attachment. A psychological study of the strange situation. Hillsdale: Lawrence-Erlbaum; 1978.
16. Salo SJ, Flykt M, Mäkelä J, Biringen Z, Kalland M, Pajulo M, et al. The effectiveness of Nurture and Play: a mentalisation-based parenting group intervention for prenatally depressed mothers. Primary health care research & development. 2019;20.

Method Design

The study consists of:

1. A randomized controlled pilot study (n=20 women/couples) carried out according to the Standard Protocol Items: Recommendations for Interventional Trials SPIRIT statement for clinical trials. The parents who agree to participate in the study will be randomly assigned in a 1:1 ratio to either the intervention or the control group, using random permuted block randomization. The participants will be informed about which group they enter at their first midwife consultation.
2. A qualitative descriptive interview study aiming to evaluate the participants' and professionals´ experience of the intervention.

Data

Data will be collected through:

* Online Questionnaires. At baseline and follow-up after the intervention, the questionnaires will be distributed to all participants through the REDcap program, regardless of whether they are in the intervention or control group. Since this is a pilot study, the study is not powered to assess effectiveness. The questionnaire data are exploratory outcomes, with a focus on identifying any potential trends. Descriptive analysis will be performed on this data. Having a control group to complete the same questionnaires as the intervention group, it is possible to compare data between the two groups, and thus identify potential trends.
* Interviews. All participants in the intervention group will be invited to an initial Parent Development Interview (PDI) to assess reflective functioning (RF). RF is an operationalization of the concept of mentalization, allowing for the evaluation of a parent´s explicit level of mentalization. The interview, coding, and analysis will be conducted by a psychologist who is trained and experienced in administering PDI interviews.
* Interviews. Some (n=15) of the participants in the intervention group will be invited to an interview about their experience of the intervention. All healthcare professionals will be invited to an interview about their experience with the intervention, including the collaboration between the hospitals and the municipality. The interviews will be performed online, by phone, in the participants' homes or at the hospital - according to the participant's preferences. Data will be analyzed using Reflexive thematic analysis by Braun and Clark, 2019.
* Videotaped settings. Emotional availability (EA): Prenatal and infancy versions observations of emotional availability (will be the primary outcome if a larger RCT will be conducted) will be conducted on semi-structured videotaped setting designed by Ann Jernberg and her colleagues called the Marschak Interaction Method (MIM). Using the MIMs, the mother (parents) is asked to perform playful activities with the fetus (Prenatal) and with their baby (postpartum) to assess Emotional availability Reflective functioning. The videotaped situation lasts about 15-20 min. EA scales are used to score the observations from the MIM setting. In the 4th edition of the original scales, EA is comprised of six dimensions - parental sensitivity, structuring, non-intrusiveness, non-hostility, child responsiveness and child involvement - rated on a seven-point Likert-type scales. All of the dimensions are rated as global perceptions (a Likert scale from 1 to 7) to capture the emotional connection in the dyad. The coding and the analysis will be carried out by a psychologist who is trained and experienced in working with EAS.

Data from medical records To identify relevant participants due to the inclusion criteria (see below), the investigators will use information from 1) the pregnancy record, where the general practitioner sends information about the pregnant women´s previous or current mental disorders to the hospital and 2) patient-reported information (PRO schema) where the pregnant women can give information about current or previous mental disorders through an electronic questionnaire. The medical records data used to identify the women will be name, CPR number, and history of mental health problems. See below for more information about the procedure.

Data from medical records will only be used by the midwives to identify relevant participants. Data from the women's medical records will thus not be forwarded to or included in any way in the project, just as no information will be obtained from the women's medical records later in the project. The only information that will be forwarded from the midwife to the project is the name and contact information (e-mail and phone number) of those who consent to hear more about the project (see below for more information about the recruitment procedure. All data included in the project will therefore solely be collected using the methods described above (see data)

Statistics In the pilot study, the aim is not to evaluate the effect. However, the investigators have made a sample size calculation for the full-scale trial. In the original effect study of the NnP, a large effect size of 1.21 was found. Contrary to the original study, the control group in our study will receive care as usual for pregnant women in a vulnerable position. the investigators therefore expect only to see medium effect sizes. A power calculation for the primary outcome measure EAS shows that using a two-sided t-test setting the significance level to 5%, estimating an effect size of 0.5 and with 80% power, we will need a sample size of N = 128, with 64 families in each group. Expecting a 20% dropout rate, the investigators will need to recruit 152 families, with 76 families in each group. Given the number of women with psychosocial vulnerabilities and estimating that around 60% will be willing to participate, it seems realistic to recruit 152 for the full-scale trial.

Descriptive statistics will be used to present categorical (n/%) and continuous variables (means (SD)). To detect differences between groups in the categorical variables, Pearson´s Chi-square test or Fischer´s exact T-test will be performed, while independent samples T-test and Mann Whitney U test will be used in the continuous variables. Missing data will be taken care of, e.g., using imputation.

Participants Inclusion criteria Pregnant women are eligible to participate in the RCT if they: 1) Have depression and/or anxiety within the previous ten years, and/or 2) use antidepressants three months prior to or during pregnancy, and/or 3) have a score of ≥11 on the Edinburg Antenatal depression Scale and/or 4) have social issues leading to antenatal care level 3 . Their partners are invited to participate, but it is not mandatory for them to participate, meaning that the women can participate without their partners if they do not wish to be part of the project. If partners participate, they do so on equal terms with the woman. This means they take part in the same activities as the pregnant women, whether they are in the intervention group or the control group.

Additional inclusion criteria for both parents: ≥18 years of age, sufficient Danish language skills to participate in NnP groups, singleton pregnancy.

Exclusion criteria Exclusion criteria for both parents include: Severe mental health disorders (e.g. schizophrenia, bipolar disorder), the child is expected to be born with a known disease, families where the infant is placed or planned placed in foster care, and families where one or both parents have an extensive use of drugs and/or alcohol. Regardless of whether this information appears in the pregnancy record, the parents will be asked about it by their midwife during the recruitment process (for more information about this process see below).

Involvement of the child As the intervention will initiate during pregnancy and continue into the postnatal period until the infant is seven months old - a period in life that is especially important for the attachment between parent and child - the study involves the newborn child (until the age of approximately 7 months). As described above (background) the parents will, among other things, be supported by healthcare professionals in their ability to read and respond appropriately to the child's emotional signals and enhance their emotional availability and attachment through caring and play activities, including postnatal activities such as baby massage, blanket swing, baby-dance, and interactive playing like peekaboo. It should be noted that the child will not be examined in any way or undergo anything other than these ordinary everyday activities. Including the child in the program is thus necessary, as the program is designed to enhance parenting abilities and the attachment between parent and child in early parenthood. The results from Finland, where the intervention, as mentioned, has been tested and is in the process of being implemented, show that involving the child brings positive outcomes, as it gives the healthcare professionals the best opportunity to provide support when they can observe the interaction between parent and child and base their guidance on concrete situations. With the aim of enhancing parenting abilities, emotional availability and attachment between parent and child, involving the child in the study significantly benefits not only the parents but also the child.

Recruitment and informed consent When referring pregnant women to Slagelse Hospital, the general practitioner informs about the pregnant women´s previous or current mental disorders. Further, the pregnant women attending Slagelse Hospital complete an electronic questionnaire at 10-12 gestational weeks, and so report information about current or previous mental disorders, social difficulties and other relevant information used to plan their antenatal care. Pregnant women fulfilling the inclusion criteria will be invited to the study together with their partner, by midwives from the hospital. When the couple come to their first midwife consultation, the midwife will give oral information about the Nurture and Play project, if the woman accepts to hear about the project. When informing the woman about the project, the midwife will clearly distinguish between what is standard antenatal care offered at the hospital and what is part of the research project.

If the woman consents to receive further information, she will be offered a choice between an informational conversation by phone or in person. She will also be informed of her right to have a support person present. Her contact information (e-mail and phone number) will be forwarded to the project team, and written information about the project, including her right to have a support person present, will be sent to her and her partner by email. The informational conversation will take place approximately 8-10 days after the initial contact, allowing her sufficient time to read the information and consider whether participating in the project is right for her. The conversation will be planned based on the woman's (and potentially her partner or other relatives) preferences regarding a phone call or in-person meeting, as well as other preferences regarding the day and time.

The informational conversation will be conducted by researcher Lotte Broberg or research assistant Frederikke Madsen, who are also midwives. At the beginning of the conversation, the woman will once again be informed of her right to have a support person present during the phone call, and if necessary, a new phone call will be arranged. During the conversation, the woman (and partner if present) will be given the opportunity to ask questions about the research project. If she, and possibly her partner, wish to participate in the project and they consent to inform their CPR number verbally, which Lotte Broberg will enter directly into REDcap, they will receive a link the consent form incl. appendix and participant information in their e-Boks via REDcap. They will be contacted again by phone within a week to make a final decision on whether they wish to participate in the project, before giving written consent online. This process gives potential participants sufficient time to consider their consent. If they decide not to participate when contacted the second time, their CPR number will no longer be stored in REDcap.

Thereafter, all the women will receive an online questionnaire assessing parental mental health, socio-demographic information, and relevant background information related to parenting. If her partner consents to participate, they will likewise receive an online questionnaire adapted to them. Finally, randomization will take place. Follow-up will take place at the end of the intervention (7 months postpartum) and consist of an online questionnaire targeted at each of the parents assessing parental mental health and the well-being of the baby, regardless of whether they are in the intervention or control group.

Regarding the child's participation in the study, informed consent will be obtained from the holder(s) of parental authority for the child, who consent on behalf of the child for him/her to participate in the project once the child is born.

The intervention group - The Nurture and Play group program In addition to care-as-usual, the intervention group will be offered to participate in the NnP adapted to include partners. The intervention consists of 11 sessions and will be provided to parents in the intervention group from around pregnancy week 26 until the child is around seven months old. Each group will consist of four to five mothers/couples. The intervention will be delivered by midwives, health nurses, and psychologists who will receive training in conducting the program. The training for the professionals will be delivered by the Finish group which has developed the program and consists of four days of training - two days introductory and two days of training that will be given after some practice with the program.

The control group - Care as Usual Existing practice for pregnant women with complex psychosocial vulnerabilities at Slagelse Hospital will be offered to women in both the intervention group and the control group. The perinatal care is guided by national guidelines from The Danish Health Authority. An extensive level of universal support from general practitioners and midwives during pregnancy and from health visitors to families with newborns during their first year of life is recommended. All pregnant women are offered a basic package of antenatal care consisting of three consultations with their general practitioner, two ultrasound examinations, and four to seven consultations with midwives depending on parity. Postnatal examinations of the infant are performed regularly by the health nurse in the infant's home, including measuring growth and evaluating the infant's physical and emotional development. During the child's first year, the health visitor examines the infant at least twice within the first three weeks after birth, at two months, at four months (for first-time mothers) and again at eight months. Extra counselling home visits to vulnerable families after the infant is born are provided by health visitors in all municipalities with the number and content depending on families' specific needs. To avoid transmission of the intervention to the control group, participants from the control group will receive visits from health nurses not trained in providing the NnP. Number of consultations with midwives, visits from health nurses and other provided perinatal services will be monitored for all participants.

Ethics It is a group of pregnant women in a vulnerable position, but a group the investigators already intend to offer extended antenatal care. Often more frequent and lengthier consultations. There is a potential risk that the participation may reopen old traumas, but the professionals are trained to handle this, ensuring that none of the participants are left alone with difficult emotions. Further, there is already positive experience with this intervention, it has been tested, evaluated, and in the process of being implemented elsewhere.

The results from the study will provide needed knowledge about the perinatal group-based family intervention in the parenting of women with psychosocial vulnerabilities. Therefor the results can be used to guide the future planning and organization of perinatal care on how to support parenting already before the child is born. Thus, the study not only benefits the participants but, to a great extent also, future parents.

By this the project will build up capacity within the perinatal mental health research environment in Denmark. Finally, the study will be one of the first Danish studies to pilot-test a group-based perinatal parenting intervention for women with psychosocial difficulties and their partners.

Risks The intervention has been tested in Finland, with no negative consequences reported, but only positive outcomes, such as reducing the depressive symptoms in parents that can otherwise complicate parenting ability, as well as emotional availability and attachment between parent and child. Based on this, the investigators therefore find the project ethically responsible and the investigators does not expect that there will be negative side effects from participating in the research project for either the parents or the child. On the opposite, by participating in the project, parents will have an even greater opportunity to receive specialized and individualized help and support during pregnancy and early parenthood from relevant professionals than what is offered in the extended antenatal care program. The therapeutic benefit of participating in the project is therefore significant.

However, there may be unforeseen risks or burdens with the intervention that the investigators are not aware of. If unforeseen conditions arise during pregnancy or childbirth, the investigators will assess whether it is necessary to interrupt the course of the research project. The trial is covered by patient insurance.

Regulation and data protection The data protection regulation and the data protection law will be obeyed. The project has been Registered in the Capital Region of Denmark's research registry, Privacy, p-2024-17353.

Economy It is midwife and ass. Prof, KU, Lotte Broberg, who has initiated the study that is anchored at Slagelse Hospital in close collaboration with the Section for Intersectoral Health Services Research, Center for Clinical Research and Prevention, The Danish Capital Region, the municipality of Slagelse (health nurses, psychologists and family therapists), as well as the Department of Psychology, University of Copenhagen. Representatives from the psychiatric healthcare services in the Region Zealand will be invited to participate in the project.

The study will be organized with a project group and a research team. The project group will consist of professionals from the participating organizations and the research project manager. The research team will consist of Head of section, and senior scientific researcher Michaela Schiøtz from Center for Clinical Research and Prevention; RM, ass. Prof. Lotte Broberg, in a joint position between Center for Clinical Research and Prevention and Slagelse Hospital; and researcher and assistant professor Katrine Røhder, the Department of Psychology, University of Copenhagen. Michaela Schiøtz, Lotte Broberg, and Katrine Røhder were all certified in the NnP intervention in March 2023.

The study is fully funded by Region Zealands Health Research Foundation, kr. 519.969. Therefore, no additional financial support will be sought for the project. The foundation will support compensation of the staff performing the intervention and expenses for the online course Nurture and Play.

The support is paid directly to the Department of Gynecology and Obstetrics, Slagelse Hospital (konto nr. 8056376000). The research team has no financial connection to Region Zealands Health Research Foundation or other stakeholders in the trial.

The participants will not receive any compensation and/or other benefits, besides the therapeutic benefit of participating in the intervention.

Communication plan Positive, negative, and inconclusive results will be published through scientific publications and presentations in relevant forums.

ELIGIBILITY:
Inclusion Criteria:

* Known with a current or previous history of anxiety and/or depression
* Referred for labour at Slagelse Hospital

Exclusion Criteria:

* Age under 18 years old
* A need for an interpreter
* Expecting more than one child
* Known with schizophrenia or other serious mental illness
* Expecting a child with a known illness
* A history of alcohol or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2026-10-15 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
The feasibility of the NnP including both parents (The recruitment procedure and the adherence to the intervention) | 1 year
  How is the intervention or service being delivered? Is it being delivered as intended? How does the actual delivery of the intervention or service differ from what was initially expected? What factors influence delivery and how? What are the difficulties faced in delivery? What are practitioners' experiences of delivering the intervention? What are the perceived supporting factors or barriers to effective delivery? How successful, or not, has it been at recruiting participants and why? Has the recruitment strategy been successful in reaching intended participants for the intervention? How successful or not has it been at retaining participants, and why? Did the participants find the intervention engaging and useful? To what extent has it reached its intended audience?
The participant's and professional´s experience of the intervention as well as the collaboration between the hospitals and the municipalities. | Approximately 30 minutes per interview
  Interviews. The interviews will be performed online, by phone, in the participants' homes or at the hospital - according to the participant's preferences. Data will be analyzed using Reflexive thematic analysis by Braun and Clark, 2019.

CONTACTS AND LOCATIONS:
Overall Officials: Michaela Schiøtz, PhD, Study Director — Bispebjerg og Frederiksberg Hospitaler

IPD SHARING:
Plan to Share IPD: No